CLINICAL TRIAL: NCT02662907
Title: Cough, Expiratory Training, and Chronic Aspiration After Head and Neck Radiotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: IRG (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0238; NCI-2016-00174 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-01-14; First posted 2016-01-26 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Post-radiotherapy H&N cancer survivors; Aspiration; Expiratory muscle strength training; EMST; Dysphagia therapy; Modified barium swallow; Neurocognitive exams; Questionnaires; Surveys; Digital Manometer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires; Barium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Aspirators Group (Experimental): Participants receive modified barium swallow at baseline and after 8 weeks of using the expiratory muscle strength training (EMST) device. Participants given neurocognitive exams at baseline. Questionnaires completed about symptoms and quality of life at baseline, after 8 weeks of using the EMST device, and 12 months after completing the study.
  Participant uses the EMST device at home on a 5-5-5 schedule (5 repetitions, 5 sets, 5 days per week) for 8 weeks.
  Digital manometer used to test how forcefully participant is able to exhale and cough at baseline, and one time each week for 8 weeks while using the EMST device.
  Interventions: Procedure: Barium Swallow; Behavioral: Questionnaires; Device: Expiratory Muscle Strength Training (EMST) Device; Device: Digital Manometer; Behavioral: Neurocognitive Exams; Drug: Barium
- Non-Aspirators Group (Other): Participants receive modified barium swallow at baseline. Participants given neurocognitive exams at baseline. Questionnaires completed about symptoms and quality of life at baseline and at 12 months.
  Interventions: Procedure: Barium Swallow; Behavioral: Questionnaires; Behavioral: Neurocognitive Exams; Drug: Barium

INTERVENTIONS:
Procedure: Barium Swallow — Participants receive modified barium swallow at baseline and after 8 weeks of using the EMST device
Behavioral: Questionnaires — Questionnaires completed about symptoms and quality of life at baseline, after 8 weeks of using the EMST device, and 12 months after completing the study.
  Other Names: Surveys
Device: Expiratory Muscle Strength Training (EMST) Device — Participant uses the EMST device at home on a 5-5-5 schedule (5 repetitions, 5 sets, 5 days per week) for 8 weeks.
  Other Names: EMST
  Arms: Aspirators Group
Device: Digital Manometer — Digital manometer used to test how forcefully participant is able to exhale and cough at baseline, and one time each week for 8 weeks while using the EMST device.
  Arms: Aspirators Group
Behavioral: Neurocognitive Exams — Participants given neurocognitive exams at baseline.
Drug: Barium — Participants receive barium prior to modified barium swallow at baseline and after 8 weeks of using the EMST device.

SUMMARY:
The goal of this clinical research study is to learn if exercising the muscles that help you cough and swallow, called expiratory muscle strength training (EMST), can help reduce the risk of pneumonia due to aspiration (inhaling saliva instead of swallowing it) in patients who have had radiation for head and neck cancer.

DETAILED DESCRIPTION:
Study Visits:

If you are found to be eligible and you agree to take part in the therapeutic portion of the EMST therapy study, you will be trained how to use the EMST device. This device is designed to help strengthen the muscles used for swallowing and coughing. To use this small handheld device, you will wear a nose clip to prevent air from coming out of your nose. You will be asked to sit upright and take a deep breath, hold your breath for a moment, and then blow forcefully into the device until you break the seal.

You will use the EMST device at home on a 5-5-5 schedule (5 repetitions, 5 sets, 5 days per week) for 8 weeks. Using the EMST device should take about 15 minutes each day you train.

One (1) time each week during these 8 weeks, you will meet with a speech pathologist in the Head and Neck Center at MD Anderson. At each visit, you will use the digital manometer to re-test how forcefully you are able to exhale and cough. The resistance of the EMST device will be adjusted based on each week's measurement.

Length of Study:

You will be on study for up to 12 months. Your study participation will be over after the follow-up call, described below. You will be taken off study early if you are unable to use the EMST device, if the doctor thinks it is in your best interest, or if you are unable to follow study directions.

Follow-Up Visit:

After 8 weeks of using the EMST device, you will have a follow-up visit.

* You will have the same functional testing you had at screening (the modified barium swallow and tests of your tongue strength, mouth opening, and ability to exhale and cough forcefully).
* You will complete the questionnaires and will be asked about your symptoms and quality of life.

Follow-Up Call:

You will be contacted by phone 12 months after you joined the study to complete 4 questionnaires about your symptoms, health and quality of life. This call should take up to 15 minutes.

This is an investigational study. The EMST device is FDA approved for exercising the muscles used in coughing and swallowing. Its use in preventing aspiration in patients who have received radiation for head and neck cancer is considered investigational.

Up to 300 patients will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years
2. History of curative-intent radiotherapy at MDACC for a new primary H&N cancer in past 15 years
3. Referred to Section of Speech Pathology and Audiology for swallowing evaluation
4. Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

1. History of recurrent or second primary H&N, central nervous system, or thoracic cancer at time of modified barium swallow (MBS) study
2. Prior H&N surgery excluding diagnostic procedures, transoral surgery, or non-radical neck dissection
3. History of functionally limiting chronic or acute cardiac, pulmonary, or neuromuscular disease
4. Tracheotomy or oxygen dependence at time of MBS
5. Patients with Mini-Mental State Examination (MMSE) <24 will be ineligible for participation in the therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Association Between Aspiration and Expiratory Function Using Expiratory Training in Post-Radiotherapy H&N Cancer Survivors | 12 months
  Primary analysis is association between baseline Penetration-Aspiration Scale (PAS) scores and baseline maximum expiratory pressures (MEPs). Analysis examined by plotting the data and computing a polyserial correlation coefficient. Participants with PAS≥6 coded as aspirators.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A. Hutcheson, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org